CLINICAL TRIAL: NCT04047836
Title: Vaping High vs. Low Nicotine E-Liquid
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Please see NCT04053868 for the current version of this study
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 19-27571; 5R01DA031193 (NIH)
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Risk Factor; Nicotine Dependence
Keywords: E-Cigarettes; Vaping; E-Cig Mods; E-Liquid
MeSH Terms: conditions — Tobacco Use Disorder; Vaping | interventions — Culture Media

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Nicotine (Other): Using an electronic cigarette, the patient will participate in a standardized vaping session using 3 mg/ml nicotine e-liquid.
  Interventions: Other: Low Nicotine E-Liquid
- Medium or High Nicotine (Other): The patient will participate in a standardized vaping session using either an electronic cigarette with 18 mg/ml nicotine e-liquid or a JUUL device with a JUUL e-liquid pod.
  Interventions: Other: Medium or High Nicotine E-Liquid

INTERVENTIONS:
Other: Low Nicotine E-Liquid — Participants will vape e-liquid with nicotine concentration of 3 mg/ml.
  Arms: Low Nicotine
Other: Medium or High Nicotine E-Liquid — Participants will vape either e-liquid with nicotine concentration of 18 mg/ml or a JUUL device with JUUL pod of 59 mg/ml nicotine e-liquid.
  Arms: Medium or High Nicotine

SUMMARY:
This study will examine the effects of electronic cigarette e-liquid nicotine content in a randomized, crossover clinical and behavioral pharmacology study of experienced adult e-cigarette users (N=36). The specific aim is to determine the impact of nicotine content of e-liquid on nicotine pharmacology, systemic exposure to toxic volatile organic compounds, and short-term cardiovascular effects.

DETAILED DESCRIPTION:
This is a within-subjects, crossover design of advanced electronic cigarette users in which we will examine nicotine pharmacokinetics, subjective effects, daily nicotine intake and nicotine titration, short-term cardiovascular effects, and toxicant exposure when participants are using low vs. high nicotine e-liquids.

Hypothesis 1: E-cigarette users will titrate their intake of nicotine such that they will inhale fewer aerosol toxicants and suffer less harm to health when using higher vs. lower nicotine content e-liquids.

Hypothesis 2: Compared to low nicotine, high nicotine e-liquid use will have similar cardiovascular effects throughout the day (due to compensatory behavioral changes), with similar effects on heart rate, blood pressure, and catecholamine release.

Hypothesis 3: Exposure to volatile organic compounds (VOCs) will be lower when vaping high nicotine e-liquids compared to low nicotine e-liquids.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of medical history and limited physical examination, as described below:
* Heart rate < 105 beats per minute (BPM)*
* Systolic Blood Pressure < 160 and > 90*
* Diastolic Blood Pressure < 100 and > 50*

  *Considered out of range if both machine and manual readings are above/below these thresholds.
* Age: >= 21 years
* Age: <= 70 years
* Current regular user of open tank electronic cigarette (EC) (at least 20 times in the past 30 days) with e-liquid nicotine of 3-6 mg/mL.
* Non-smoker or non-daily cigarette smokers agreeing to abstain from cigarettes for the duration of the study.
* Saliva cotinine >50 ng/mL and/or NicAlert=6
* Carbon monoxide >= 5 ppm or per discretion of Principal Investigator

Exclusion Criteria:

* Medical
* Heart disease
* Seizures
* Cancer
* Thyroid disease (okay if controlled with medication)
* Diabetes
* Hepatitis B or C or Liver disease
* Glaucoma
* Kidney disease or urinary retention
* History of stroke
* An ulcer in the past year
* Active use of an inhaler for Asthma or Chronic obstructive pulmonary disease (COPD)
* Psychiatric conditions
* Current or past schizophrenia, and/or current or past bipolar disorder
* Major depression, current or within the past year
* Major personality disorder
* Participants with current or past minor or moderate depression and/or anxiety disorders will be reviewed by the PI and considered for inclusion
* History of psychiatric hospitalizations is not exclusionary, but study participation will be determined as per PI's approval
* Drug/Alcohol Dependence
* Alcohol or illicit drug dependence within the past 12 months with the exception of those who have recently completed an alcohol/drug treatment program
* Positive toxicology test for illicit drugs at the screening visit (THC & prescribed medications okay)
* Opioid replacement therapy (including methadone, buprenorphine, or other)
* Psychiatric medications
* Current regular use of any psychiatric medications with the exception of Selective Serotonin Reuptake Inhibitors (SSRIs) and serotonin-norepinephrine reuptake Inhibitors (SNRIs) and current evaluation by the PI that the participant is otherwise healthy, stable, and able to participate.
* Medications
* Use of medications that are inducers of nicotine metabolizing enzyme CYP2A6 (Example: rifampicin, carbamazepine, phenobarbital, and other anticonvulsant drugs).
* Use of sympatholytic medications for cardiovascular conditions including hypertension (Example: beta and alpha-blockers)
* Concurrent use of nicotine-containing medications
* Any stimulant medications (example: Adderall) generally given for attention deficit hyperactivity disorder (ADHD) treatment
* Other/Misc. Chronic Health Conditions
* Oral thrush
* Fainting (within the last 30 days)
* Other "life threatening illnesses" as per PI's discretion
* Pregnancy
* Pregnancy (self-reported and urine pregnancy test)
* Breastfeeding (determined by self-report)
* Concurrent participation in another clinical trial
* Inability to read and write in English
* Planning to quit vaping within the next 60 days
* Concurrent regular use of marijuana (occasional users of these products may be enrolled if they agree to abstain from their use during the period of the study)
* Use of other tobacco products, smokeless tobacco, pipes, cigars/cigarillos, blunts/spliffs (no more than 10 times in the past month and must agree to abstain from their use during the period of the study)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Nicotine Exposure | Day 1 of each Arm
  Plasma nicotine area under curve (AUC) (ng/ml*h)
Cardiovascular Effects: Heart Rate | Days 1-3 of each Arm
  Participant heart rate will be measured in beats per minute throughout the inpatient stay.
Cardiovascular Effects: Systolic Blood Pressure | Day 2 of each Arm
  Participant systolic blood pressure will be taken for 24 hours during ad-lib e-cigarette use.
Cardiovascular Effects: Diastolic Blood Pressure | Day 2 of each Arm
  Participant diastolic blood pressure will be taken for 24 hours during ad-lib e-cigarette use.

SECONDARY OUTCOMES:
Vaping Topography: Puff Number | Days 1-3 of each Arm
  Vaping topography measures will be obtained from self-reported participant vaping log during the ad libitum sessions and measured as puffs per minute.
Vaping Topography: Puff Duration | Days 1-3 of each Arm
  Vaping topography measures will be obtained from self-reported participant vaping log during the ad libitum sessions and measured as seconds per puff.
Vaping Topography: Inter-Puff Interval | Days 1-3 of each Arm
  Vaping topography measures will be obtained from self-reported participant vaping log during the ad libitum sessions and measured as seconds/minutes between puffs.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Benowitz, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California

IPD SHARING:
Plan to Share IPD: No